CLINICAL TRIAL: NCT01911390
Title: Effect of Rice Bran and Cooked Navy Beans on Cholesterol Levels in Healthy Children Involved in the Healthy Hearts Program
Brief Title: Effect of Rice Bran and Cooked Navy Beans on Cholesterol Levels in Healthy Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Poudre Valley Health System (Other)
Collaborators: Colorado State University (Other)
Responsible Party: Principal Investigator, Gary J. Luckasen, MD, Co-Principal Investigator, Poudre Valley Health System
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Version 06/18/2013
Record Dates: First submitted 2013-07-25; First posted 2013-07-30 (Estimated); Results first posted 2017-04-05 (Actual); Last update posted 2017-05-15 (Actual); Status verified 2017-05

CONDITIONS: Hyperlipidemias
Keywords: High cholesterol.
MeSH Terms: conditions — Hyperlipidemias; Hypercholesterolemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Control Arm (Placebo Comparator): No bean or rice bran additive in smoothie or muffin.
  Interventions: Dietary Supplement: Control arm
- Bean powder (Active Comparator): 1/4 cup beans (17.5 grams powder)/day in smoothie or muffin.
  Interventions: Dietary Supplement: Bean powder
- Rice bran (Active Comparator): 15 grams rice bran/day in smoothie or muffin.
  Interventions: Dietary Supplement: Rice bran
- Bean powder and rice bran (Active Comparator): 9 grams bean powder/day and 8 grams rice bran /day in smoothie or muffin.
  Interventions: Dietary Supplement: Bean powder and rice bran

INTERVENTIONS:
Dietary Supplement: Bean powder — Archer Daniels Midland (ADM) Edible Bean Specialties, Inc. will supply cooked navy bean powders.
  Arms: Bean powder
Dietary Supplement: Rice bran — USDA (Beaumont, TX) provided rice bran for meals that was polished from U.S. rice mills using U.S. grown rice varieties.
  Arms: Rice bran
Dietary Supplement: Control arm — No bean or rice bran additive in smoothie or muffin.
  Other Names: Placebo Comparator
  Arms: Control Arm
Dietary Supplement: Bean powder and rice bran — Archer Daniels Midland (ADM) Edible Bean Specialties, Inc. will supply cooked navy bean powders. USDA (Beaumont, TX) provided rice bran for meals that was polished from U.S. rice mills using U.S. grown rice varieties.
  Other Names: Bean Powder & Rice Bran
  Arms: Bean powder and rice bran

SUMMARY:
A multidisciplinary team of clinicians and researchers will conduct a pilot feasibility study to evaluate whether dietary intake of dry bean powder or rice bran or a combination is a helpful dietary recommendation to reduce total cholesterol levels in children with identified, modifiable CVD risk factors, elevated total cholesterol and obesity. Consumption of dry bean powder and rice bran merit additional investigation to study feasibility and acceptability in children and how they influence their lipid levels or obesity.

DETAILED DESCRIPTION:
Children will be screened prior to participation with the expectation of enrolling 40 to randomize equally to either the control arm or one of the three intervention arms. This should assure that at least 10 participants would complete each intervention. The four groups are placebo (no bean powder or rice bran included), 1/4 cup cooked navy bean powder (17.5grams powder)/day, 15 grams rice bran/day, and combination of 9 grams of bean powder/day and 8 grams rice bran/day. Participants will follow this dietary intervention by being provided a study snack, such as a banana nut muffin and strawberry-pineapple smoothie. Participants will consume one snack on a daily basis for a total of four weeks (28 days). The snack options were developed by a professional chef and research dietitian to fit a set of requirements for calorie and macronutrient content based on USDA food guide recommendations. The placebo group will be provided the same snacks without the inclusion of rice bran or bean powder.

Randomization of subjects to the dietary intervention groups will be done during the study enrollment period. Randomization will be based on sex of the subject to include equal numbers of both genders across all 4 groups.

All participants will consume the allocated foods daily for a total of four weeks (28 days) and will not be required to alter the rest of their diets in any other way. They will also complete a 3-day food and activity log each week, starting the week prior to the study intervention (Week 0) and ending the week of their final visit (Week 4).

ELIGIBILITY:
Inclusion Criteria:

* Children between the ages of 8-13 years old who were screened by the Healthy Hearts Club
* Non-fasting total cholesterol greater than or equal to 180 mg/dl
* Non-fasting LDL greater than or equal to 100mg/dl
* Non-fasting HDL less than 60mg/dl
* Willing to consume study provided ingredient (cooked dry bean powder or rice bran or combination) for 28 consecutive days.

Exclusion Criteria:

* History of food allergies and/or major dietary restrictions
* Taking prescribed medication
* Ongoing medical illness

Ages: 8 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 41 (Actual)
Dates: Start 2013-07 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Ryan, PhD, Principal Investigator — Colorado State University; Gary Luckasen, MD, Principal Investigator — University of Colorado Health
Locations (2):
- United States (2):
  - Colorado State University, Fort Collins, Colorado
  - Medical Center of the Rockies, Loveland, Colorado

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Li KJ, Borresen EC, Jenkins-Puccetti N, Luckasen G, Ryan EP. Navy Bean and Rice Bran Intake Alters the Plasma Metabolome of Children at Risk for Cardiovascular Disease. Front Nutr. 2018 Jan 19;4:71. doi: 10.3389/fnut.2017.00071. eCollection 2017. PMID 29404331

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study proposed to randomize approximately 40 subjects to complete 38.
Pre-assignment Details: A total of 41 subjects were screened and assented. Of the subjects assessed, 38 (93%) completed the trial with 3 (7%) withdrawn for noncompliance of required food consumption.
Period: Overall Study
Arm/Group | Control Arm | Bean Powder | Rice Bran | Bean Powder and Rice Bran
Started | 10 | 10 | 10 | 11
Completed | 9 | 10 | 9 | 10
Not Completed | 1 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Children aged 8-13 years old at risk for CVD due to abnormal lipids were recruited. Elevated cholesterol levels were defined as total cholesterol ≥180mg/dL and HDL <60mg/dL; LDL ≥100mg/dL and HDL <60mg/dL; or non-HDL >100mg/dL and HDL <60mg/dL.
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Arm | Bean Powder | Rice Bran | Bean Powder and Rice Bran | Total
Number analyzed (Participants) | 10 | 10 | 10 | 11 | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 10 (1) | 10 (1) | 10 (1) | 10 (1) | 10 (1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 6 | 5 | 20
  Male | 6 | 5 | 4 | 6 | 21
Region of Enrollment [Number; unit: participants]
  United States | 9 | 10 | 9 | 10 | 38

OUTCOME MEASURES:

1. Primary Outcome: Total Cholesterol
Description: The primary outcome variable to be studied is total cholesterol. A full lipid panel report will also provide information on LDL, HDL, triglycerides etc.
Time Frame: Baseline, 4 weeks
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Control Arm | Bean Powder | Rice Bran | Bean Powder and Rice Bran
Number analyzed (Participants) | 9 | 10 | 9 | 10
mg/dL
  Baseline Tchol Average | 166 (13) | 178 (30) | 167 (16) | 169 (26)
  4 week post Tchol Average | 165 (20) | 172 (33) | 171 (18) | 168 (22)

2. Secondary Outcome: Palatability
Description: Other outcomes include palatability and acceptability of study-provided snacks that include cooked navy bean powder, rice bran, or a combination in children. The participants will fill out questionaires describing how the products tasted and how much they consumed.
Time Frame: Baseline, 4 weeks
Population: The criteria used to quantify GI discomforts or issues included participants who responded 'yes' to any GI discomfort and rated the discomfort level ≥3 out of a 5-point scale.
Measure: Count of Participants; unit: Participants
Arm/Group | Control Arm | Bean Powder | Rice Bran | Bean Powder and Rice Bran
Number analyzed (Participants) | 9 | 10 | 9 | 10
Participants | 3 | 1 | 3 | 1

ADVERSE EVENTS:
Arm/Group | Control Arm | Bean Powder | Rice Bran | Bean Powder and Rice Bran
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/10 | 0/9 | 0/10
Other Adverse Events (participants affected / at risk) | 0/9 | 0/10 | 0/9 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No